CLINICAL TRIAL: NCT04303598
Title: A Randomized, Double-blind, Double-simulated, Active-controlled，Phase III Clinical Study Evaluating the Efficacy and Safety of Azvudine Combined With Tenofovir Fumarate and Efavirenz in Hiv-infected Treatment Naive Patients
Brief Title: Phase III Clinical Study of Azvudine in Hiv-infected Treatment Naive Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GQ-FNC-301
Record Dates: First submitted 2020-03-04; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: HIV-infection/Aids
Keywords: FNC; HIV-infection; Aids
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — azvudine; Lamivudine; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The experiment was conducted under a randomized method, each center disputed into the group via competition. Treatment assignment was carried out in accordance with a central randomization schedule generated with SAS (version 9.4). Randomization was done by a computer-generated system (IWRS). The randomization table (1st blind code) and second blind code were sealed and stored in triplicate offices of the sponsor, investigator and the independent statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FNC Treatment Group (Experimental): FNC 3mg, 1 tablet;TDF 300mg, 1 tablet;EFV 200mg, 2 tablets;3TC placebo 1 tablet;daily oral before bedtime
  Interventions: Drug: FNC; Drug: TDF; Drug: EFV; Drug: 3TC placebo
- 3TC control group (Active Comparator): 3TC 300mg, 1 tablet;TDF 300mg, 1 tablet;EFV 200mg, 2 tablets;FNC placebo 1 tablet;daily oral before bedtime
  Interventions: Drug: 3TC; Drug: TDF; Drug: EFV; Drug: FNC placebo

INTERVENTIONS:
Drug: FNC — 3mg, 1 tablet，QD
  Other Names: Azvudine
  Arms: FNC Treatment Group
Drug: 3TC — 300mg, 1 tablet，QD
  Other Names: Lamivudine
  Arms: 3TC control group
Drug: TDF — 300mg, 1 tablet，QD
  Other Names: Tenofovir Fumarate
Drug: EFV — 200mg, 1 tablet，QD
  Other Names: Efavirenz
Drug: FNC placebo — 1 tablet，QD
  Other Names: Azvudine placebo
  Arms: 3TC control group
Drug: 3TC placebo — 1 tablet，QD
  Other Names: Lamivudine placebo
  Arms: FNC Treatment Group

SUMMARY:
Azvudine,(FNC)， new nuclear nucleoside reverse transcriptase inhibitors, FNC make itself a better candidate to be co-formulated in other anti-HIV therapies, thus to improve patient's compliance, approved by state drug administration (NMPA) for clinical research. FNC has completed its phase I、II clinical studies with desirable results.This is a multi-center, randomized, double-blind,double-placebo,active-control clinical trial. Subjects in experimental arm receives FNC+TDF+EFV+3TC placebo, while the subjected in active control arm receives 3TC+TDF+EFV+FNC placebo. The background drugs in both arms are conducted in open-label design while FNC and 3TC are conducted in double-blinded design.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old, regardless of gender;
2. Participant must have an positive HIV test;
3. Have not received anti-HIV treatment;
4. HIV-1 RNA≥1000 copies/ml and the investigators determined that the subjects were eligible for HAART therapy.
5. Who have no recent family planning and agree to take effective non-drug contraceptive measures during the trial period and within 3 months after the end of administration;
6. The subjects could fully understand the purpose, nature, method and possible adverse reactions of the test, and voluntarily participate in and sign the informed consent.

Exclusion Criteria:

1. History of allergy to any ingredient or excipient of the research drug or have a high sensitivity constitution;
2. Patients with severe opportunistic infection or tumor;
3. Clinically Hepatitis b surface antigen/hepatitis c antibody positive;
4. Clinically Alanine transaminase and/or alanine transaminase ≥5× normal upper limit (ULN);
5. Clinically Alanine aminotransferase ≥3×ULN and total bilirubin ≥2×ULN (direct bilirubin/total bilirubin > 35%);
6. Glomerular filtration rate < 70ml/min/1.73m2 (calculated by ckd-epi Creatinine 2009 Equation), or Creatinine ≥ULN;
7. Clinically significant diseases serious chronic diseases , metabolic diseases (such as diabetes), neurological and psychiatric diseases;
8. History of pancreatitis;
9. Women in pregnancy and breastfeeding;
10. History of drug abuse, alcohol abuse and drug abuse;
11. Participating in clinical trials of other drugs within the first three months of screening;
12. Other factors considered inappropriate by the investigator to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of subjects with plasma HIV-1 Ribonucleic acid (RNA) <50 copies/milliliter (c/mL) at Week 48 | 48 Weeks
  Rate of participants with a HIV-1 RNA < 50 copies per mL .If HIV RNA level is < 50 copies per mL at Week 48, it is considered as virologic success as per the snapshot approach.

SECONDARY OUTCOMES:
Rate of subjects with plasma HIV-1 Ribonucleic acid (RNA) <50 copies/milliliter (c/mL) at Week 24 and Week 96 | Week 24 and Week 96
  Rate of participants with a HIV-1 RNA < 50 copies per mL at Week 24 and Week 96
Rate of subjects with plasma HIV-1 Ribonucleic acid (RNA) <400 copies/milliliter (c/mL) at Week 24 ，Week 48 and Week 96； | Week 24 and Week 48 and Week 96,
  Rate of participants with a HIV-1 RNA < 50 copies per mL at Week 24，Week 48 and Week 96
Change of CD4+ cell count from baseline at Week 48 and Week 96 | Week 48 and Week 96
  The immunologic change was determined by changes in Cluster of CD4+ cell count. Change from baseline in CD4+ cell count at Weeks 48 and 96 were assessed
Time to achieve virologic failure（HIV-1 RNA<50 copies/ml） | Baseline and Week 96
  Time to HIV-1 RNA<50 copies/ml from baseline
Diachronic change of logarithm (log) HIV-RNA reduction from baseline | Baseline and Week 96
  The Diachronic change of logarithm (log) HIV-RNA change was determined by changes in Cluster of logarithm (log) HIV-RNA count. Change from baseline in logarithm (log) HIV-RNA at Weeks 96 were assessed
Diachronic change of CD4+T、 CD8+T cell count from baseline | Baseline and Week 96
  The immunologic change was determined by changes in Cluster of CD4+ cell count. Change from baseline in CD4+ cell count to Weeks 96 were assessed
Safety outcome of subjects at Week 48 and Week 96。 | Week 48 and Week 96
  Rate of participants discontinuing therapy due to AEs were reported. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing DiTan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Public Health Medical Center, Chongqing, Chongqing Municipality
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - Wuhan Jinyintan Hospital, Wuhan, Hebei
  - The Fouth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The First Hospital of Changsha, Changsha, Hunan
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - The Public Health Clinical Center of Chengdu, Chengdu, Sichuan
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - Xixi Hospital of Hangzhou, Hangzhou, Zhejiang